CLINICAL TRIAL: NCT02901548
Title: A Phase 2 Study of Check Point Inhibitor, Durvalumab (Medi4736) for Bacillus Calmette-Guérin (BCG) Refractory Urothelial Carcinoma in Situ (CIS) of the Bladder
Brief Title: Phase 2 Durvalumab (Medi4736) for Bacillus Calmette-Guérin (BCG) Refactory Urothelial Carcinoma in Situ of the Bladder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed early due to futility
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18788; ESR-15-11326 (Other Grant/Funding Number: AstraZeneca)
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Results first posted 2021-06-11 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Carcinoma in Situ of Bladder; Bladder Cancer
Keywords: BCG refractory CIS; Urothelial CIS of bladder; Carcinoma in situ (CIS); Bacillus Calmette-Guérin (BCG); Medi4736; Durvalumab; CIS of the bladder; Bladder cancer; BCG Vaccine; Bladder diseases; Urothelial diseases
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma in Situ; Urinary Bladder Diseases | interventions — durvalumab; Cystoscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab Plus Cystoscopy (Experimental): Durvalumab: Fixed dose level IV infusion every 4 weeks for 13 study treatment cycles/infusions over 12 months/1 year. Cystoscopy with biopsy will be performed every 3 months to monitor the treatment response during this one year of treatment phase. It will be performed every 6 months during year 2 of the surveillance phase.
  Interventions: Drug: Durvalumab; Procedure: Cystoscopy with Biopsy

INTERVENTIONS:
Drug: Durvalumab — Durvalumab will be given every 4 weeks at 1500 mg/kg IV for total of 12 months/13 doses.
  Other Names: Medi4736
Procedure: Cystoscopy with Biopsy — Cystoscopy with biopsy and transurethral resection of the bladder tumor (TURBT) (if indicated) will be performed at baseline, month 3, 6, 9, 12, 18, and 24. The month 6 and 24 cystoscopy will be done in the operating room with mapping biopsy. Rest of the cystoscopic exam with biopsy will be performed in the out-patient office setting and if clinically indicated will be repeated in the operating room. Participants will be off study if any of the biopsies document muscle invasive (T2 or above) urothelial carcinoma. Participants will also be off study if their month 6, 9, 12, 18 biopsies show persistent (month 6) or recurrent CIS or invasive (T1 or above) urothelial carcinoma. Otherwise, participants will remain on study until after the month 24 mapping biopsy.

SUMMARY:
The purpose of this study is to test if an experimental drug called Durvalumab (Medi4736) given by intravenous (IV) infusion is effective in treating carcinoma in situ (CIS) of the bladder that no longer responds to Bacillus Calmette-Guérin (BCG) and to collect information on the safety of these drugs and whether they cause any side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must have pathologically confirmed urothelial carcinoma in situ (CIS) of the bladder that meet one of the following criteria: 1. Persistence of high-grade CIS at 6 months following an adequate course of BCG; OR - 2. Stage/grade progression at 3 months after induction BCG; OR - 3. Recurrence of high-grade CIS after achieving a disease-free state (i.e., CR) following induction of an adequate course of BCG that occurs < 9 months after the last exposure to BCG; OR - 4. Persistent CIS noted on the bladder biopsies within 3 months of completing at least 2 induction BCG (minimum of five weekly instillations). An adequate course of BCG should be defined as at least one course of induction (minimum of five weekly instillations) and one maintenance (two of three instillations) in a 6 months period, with an exception for any patient with grade/stage progression after induction BCG (minimum of five weekly instillations).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Adequate organ and marrow function.
* Written informed consent and any locally required authorization (e.g., HIPAA in the USA, EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
* Females must not be pregnant, or breast feeding and must have a negative urine or serum pregnancy test within 28 days prior to treatment on day 1. Females of childbearing potential who are sexually active with a nonsterilized male partner must use a highly effective method of contraception from the time of screening, and must agree to continue using such precautions for 90 days after the final dose of Durvalumab. They must also refrain from egg cell donation for 90 days after the final dose of Durvalumab.
* Nonsterilized males who are sexually active with a female partner of childbearing potential must use a highly effective method of contraception and refrain from sperm donation from Day 1 through 90 days after receipt of the final dose of Durvalumab.

Exclusion Criteria:

* Muscle invasive (T2 or above) urothelial carcinoma or urothelial carcinoma outside the bladder.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site) or previous enrolment in the present study.
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab.
* History of another primary malignancy except for: Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence; Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; Adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ.
* Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, tyrosine kinase inhibitor, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤ 30 days prior to the first dose of study drug and within 6 weeks for nitrosourea, mitomycin C or intravesical therapy).
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* Any unresolved toxicity (CTCAE grade 2 or above) from previous anti-cancer therapy. [Potential participants with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy)].
* Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
* Active or prior documented autoimmune disease within the past 2 years. NOTE: Potential participants with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* History of primary immunodeficiency.
* History of allogeneic organ transplant.
* History of pneumonitis.
* History of hypersensitivity to durvalumab or any excipient.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any participant known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the participant to give written informed consent.
* Known history of previous clinical diagnosis of tuberculosis.
* History of leptomeningeal carcinomatosis.
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab.
* Females who are pregnant, breast-feeding or males or females of reproductive potential who are not employing an effective method of birth control.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* Uncontrolled seizures.
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2021-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jingsong Zhang, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - Mount Sinai Medical Center Miami, Miami Beach, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Durvalumab Plus Cystoscopy
Started | 17
Completed | 13
Not Completed | 4
Not completed — Withdrew after month 3 biopsy showed persistent cancer | 4

BASELINE CHARACTERISTICS:
Arm/Group | Durvalumab Plus Cystoscopy
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate at 6 Months
Description: Complete Response Rate at month six based on the week 26 mapping biopsy in BCG refractory CIS urothelial bladder cancer. The absence of CIS of bladder on the mapping biopsies after pathological review would be considered complete response to treatment.
Time Frame: 6 Months
Population: Evaluable participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab Plus Cystoscopy
Number analyzed (Participants) | 13
percentage of participants | 23.1 [5 to 53.8]

2. Secondary Outcome: Complete Response Rate at 24 Months
Description: Complete Response Rate at month 24 based on the week 104 mapping biopsy in BCG refractory CIS urothelial bladder cancer. The absence of CIS of bladder on the mapping biopsies after pathological review would be considered complete response to treatment.
Time Frame: 24 Months
Population: Evaluable participants. Study was closed early due to futility.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab Plus Cystoscopy
Number analyzed (Participants) | 13
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected from time of informed consent to 90 days after last dose of study drug. Adverse events are still being collected (one participant still on treatment).
Arm/Group | Durvalumab Plus Cystoscopy
All-Cause Mortality (participants affected / at risk) | 3/17
Serious Adverse Events (participants affected / at risk) | 5/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab Plus Cystoscopy (N=17)
Dysuria (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash muculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Cystoprstatectomy (General disorders) | 1 (1)
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Cystoprostatectomy
Stroke (Nervous system disorders) | 1 (1)
Nervous system disorders -Other (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab Plus Cystoscopy (N=17)
Investigations- Other (Investigations) | 9 (12)
INR increased (Investigations) | 3 (5)
Serum amylase increased (Investigations) | 3 (4)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
GGT increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (4)
Renal and urinary disorders - Other (Renal and urinary disorders) | 6 (7)
Cystitis noninfective (Renal and urinary disorders) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Fatigue (General disorders) | 7 (7)
Edema limbs (General disorders) | 1 (2)
Infusion related reaction (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4)
Skin and subcutaneous tissue disorders -Other (Skin and subcutaneous tissue disorders) | 2 (2)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Headache (Nervous system disorders) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Hot flashes (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (4)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (5)
Ottis externa (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Leykocytosis (Blood and lymphatic system disorders) | 1 (1)
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Eye disorders -Other (Eye disorders) | 1 (1)
Wound complications (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
All reported deaths were on post study treatment survival follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT02901548/Prot_SAP_000.pdf